CLINICAL TRIAL: NCT06315491
Title: A Randomized Phase 2 Study of CBX 12 in Subjects With Platinum Resistant or Refractory Ovarian Cancer
Brief Title: A Study of CBX 12 in Subjects With Platinum Resistant or Refractory Ovarian Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cybrexa Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBX-12-201
Record Dates: First submitted 2024-03-07; First posted 2024-03-18 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Platinum-resistant Ovarian Cancer; Refractory Ovarian Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CBX-12 - 125mg/m2 q21d (Experimental): 125mg/m2 CBX-12 administered by intravenous (IV) infusion every 21 days. Treatment will continue until there is evidence of progressive disease (PD) or development of unacceptable toxicity.
  Interventions: Drug: CBX-12
- CBX-12 - 100mg/m2 q21d (Experimental): 100mg/m2 CBX-12 administered by intravenous (IV) infusion every 21 days. Treatment will continue until there is evidence of progressive disease (PD) or development of unacceptable toxicity.
  Interventions: Drug: CBX-12

INTERVENTIONS:
Drug: CBX-12 — CBX-12 is an alphalex construct which contains exatecan as the pharmacologically active moiety.

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and efficacy of CBX-12 in female subjects with platinum resistant or refractory ovarian cancer at 2 doses; 125 mg/m2 every 21 days or 100 mg/m2 every 21 days.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically- or cytologically-diagnosed epithelial high-grade serous cancer of the ovary, fallopian tube cancer or primary peritoneum cancer that is refractory to prior therapy and must have platinum-resistant disease defined as:

  * Subjects who have received only 1 platinum-based chemotherapy regimen for at least 4 cycles of platinum must have disease progression on treatment or occurring ≤ 26 weeks after their last dose of platinum.
  * Patients who have progressed following a second course of a platinum based regimen.
  * Subjects may have up to 2 additional systemic regimens for advanced or metastatic disease. Maintenance regimens (e.g., with a PARP inhibitor or bevacizumab) are not considered separate regimens.
* Age greater than or equal to 18 years at the time of signing the informed consent form (ICF).
* Has measurable disease per RECIST 1.1.
* Has provided written informed consent.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Adequate liver, renal, hematologic, pulmonary and coagulation function.

Exclusion Criteria:

* Cytotoxic chemotherapy, biologic agent, investigational agent, or radiation therapy within 3 weeks prior to the first dose of CBX-12.
* Subjects who are currently receiving any other anticancer or investigational agent(s).
* Clinically significant intercurrent disease.
* Active human immunodeficiency virus (HIV) infection.
* Active hepatitis B or C infection.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of Subjects With Complete Response (CR) or Partial Response (PR) [Objective Response Rate (ORR)] | Randomization to progressive disease (PD) (Up to approximately 21 months)
  ORR is defined as the proportion of subjects achieving a confirmed best overall response (BOR) of CR or PR defined using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.

SECONDARY OUTCOMES:
Incidence of Subjects With Treatment Emergent Adverse Events (TEAEs) | First dose of study drug to 30-day post-dose follow up (Up to approximately 21 months)
  Safety as assessed by the incidence of treatment-emergent AEs (TEAEs).
Median Duration of Response (DoR) | Date of Initial CR or PR to PD (Up to 21 Months)
  Duration of response is the interval from the date of initial CR or PR until the first date criteria for PD is met using RECIST v1.1 criteria, or initiation of other (or additional) antitumor therapy is first reported, or death due to any cause.
Progression-Free Survival (PFS) | Randomization to PD or Date of Death (Up to 21 Months)
  PFS is defined as the time from the day of randomization to the first evidence of progression as defined by RECIST (RECIST v1.1) criteria or death from any cause.
Plasma levels of CBX-12 (AUC0-24hr) | At 1st dose of study drug (pre-dose, end of infusion (EOI), 1, 2, and 4 hours post EOI), and 10-14 days post 1st dose
  Assessment of pharmacokinetic (PK) variable AUC0-24hr
Plasma levels of CBX-12 (Cmax) | At 1st dose of study drug (pre-dose, end of infusion (EOI), 1, 2, and 4 hours post EOI), and 10-14 days post 1st dose
  Assessment of pharmacokinetic (PK) variable Cmax
Plasma levels of CBX-12 (Tmax) | At 1st dose of study drug (pre-dose, end of infusion (EOI), 1, 2, and 4 hours post EOI), and 10-14 days post 1st dose
  Assessment of pharmacokinetic (PK) variable Tmax
Plasma levels of CBX-12 (T1/2) | At 1st dose of study drug (pre-dose, end of infusion (EOI), 1, 2, and 4 hours post EOI), and 10-14 days post 1st dose
  Assessment of pharmacokinetic (PK) variable T1/2
Plasma levels of Exatecan (AUC0-24hr) | At 1st dose of study drug (pre-dose, end of infusion (EOI), 1 hour post EOI, 2 hours post EOI, 4 hours post EOI), and 10-14 days post 1st dose
  Assessment of pharmacokinetic (PK) variable AUC0-24hr
Plasma levels of Exatecan (Cmax) | At 1st dose of study drug (pre-dose, end of infusion (EOI), 1 hour post EOI, 2 hours post EOI, 4 hours post EOI), and 10-14 days post 1st dose
  Assessment of pharmacokinetic (PK) variable Cmax
Plasma levels of Exatecan (Tmax) | At 1st dose of study drug (pre-dose, end of infusion (EOI), 1 hour post EOI, 2 hours post EOI, 4 hours post EOI), and 10-14 days post 1st dose
  Assessment of pharmacokinetic (PK) variable Tmax
Plasma levels of Exatecan (T1/2) | At 1st dose of study drug (pre-dose, end of infusion (EOI), 1 hour post EOI, 2 hours post EOI, 4 hours post EOI), and 10-14 days post 1st dose
  Assessment of pharmacokinetic (PK) variable T1/2

CONTACTS AND LOCATIONS:
Overall Officials: Michael Needle, MD, Study Director — Cybrexa Therapeutics
Locations (17):
- United States (17):
  - Honor Health, Scottsdale, Arizona
  - Arizona Oncology Associates, Tucson, Arizona
  - Usc Norris Comprehensive Cancer Center, Los Angeles, California
  - Yale University School of Medicine, New Haven, Connecticut
  - D&H Cancer Research Center, Margate, Florida
  - South Florida Gynecology, Tampa, Florida
  - Northwest Cancer Centers, Dyer, Indiana
  - Norton Cancer Institute, Louisville, Kentucky
  - Women's Cancer Care, Covington, Louisiana
  - Pci Nyu Langone Health, New York, New York
  - Albert Einstein College of Medicine Montefiore Medical, New York, New York
  - University Hospitals Seidman Cancer Center, Cleveland, Ohio
  - Oncology Associates of Oregon, Eugene, Oregon
  - Allegheny Singer Research Institute D/B/A Ahn Research Institution, Pittsburgh, Pennsylvania
  - Mary Crowley Cancer Research, Dallas, Texas
  - Texas Oncology- Gulf Coast, The Woodlands, Texas
  - Multicare Institute For Research & Innovation, Tacoma, Washington